CLINICAL TRIAL: NCT05675488
Title: Ultrasound Features of Trigger Finger: A Comparative Study With Healthy Volunteers
Brief Title: Ultrasound Features of Trigger Finger
Status: Completed | Type: Observational
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Yasin Demir, Associated Proffessor, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Other Study IDs: 31
Record Dates: First submitted 2022-12-29; First posted 2023-01-09 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Trigger Finger
MeSH Terms: conditions — Trigger Finger Disorder | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Trigger Finger Patients
  Interventions: Diagnostic Test: Ultrasound
- Healthy individuals
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — Thickness of flexor tendon and A1 pulley at MCP joint level

SUMMARY:
Our aim in this study; to compare the ultrasound findings seen in trigger finger patients with healthy volunteers. Thus, ultrasound findings associated with trigger finger development will be documented

DETAILED DESCRIPTION:
A1 pulley thickness, flexor tendon thickness, and presence of nodules at the MCP joint level of the trigger finger patients will be recorded. The same measurements will be made in age- and sex-matched healthy volunteers, followed by comparison and analysis.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 years
* To have trigger finger (for patient group)
* Not to have trigger finger (for healthy group)

Exclusion Criteria:

* Aged under 18
* Wound or infection in the imaging area

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 30 patients with trigger finger and 30 age and BMI-matched healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-01-14 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-08-07 (Actual)

PRIMARY OUTCOMES:
Thickness of flexor tendon | through study completion, an average of one and a half months
  Thickness of flexor tendon at MCP joint level
Thickness of A1 pulley | through study completion, an average of one and a half months
  Thickness of A1 pulley at MCP joint level

SECONDARY OUTCOMES:
Presence of nodules | through study completion, an average of one and a half months
  Presence of nodule in flexor tendon

CONTACTS AND LOCATIONS:
Overall Officials: Yasin Demir, Principal Investigator — Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Locations (1):
- Gaziler FTR EAH, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kamaci GK, Demir Y, Okur G, Ceylan H, Cetinturk H, Artuc SE, Ekinci U, Guzelkucuk U, Aydemir K. Comparison of Ultrasonographic Features Among Healthy Individuals and Patients With Trigger Finger. J Clin Ultrasound. 2025 Sep 11. doi: 10.1002/jcu.70080. Online ahead of print. PMID 40934299